CLINICAL TRIAL: NCT05749120
Title: Recipient Vessels for Free Tissue Flaps in Advanced Oncologic Defects of the Midface and Scalp: Prospective Randomized Study
Brief Title: Recipient Vessels for Free Tissue Flaps in Advanced Oncologic Defects of the Midface and Scalp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Principal Investigator, Bruno Albuquerque, MD, Principal investigator, Instituto Nacional de Cancer, Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 89042418.7.0000.5274
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Head Neck Neoplasms
Keywords: microanastomosis; free tissue flaps; cervical vessels; superficial temporal vessels; advanced reconstruction
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel group trial design with allocation ratio of 1:1 and permuted block randomization
Who Masked: Participant
Masking Description: The care provider knows the surgical intervention and the randomized participant doesn´t know the recipient vessel performed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superficial temporal recipient vessels (group A) (Experimental): Participants in whom superficial temporal vessels were used as the recipient vessels.
  Interventions: Procedure: Recipient vessel selected for microanastomosis
- Cervical recipient vessels (group B) (Active Comparator): Participants in whom cervical vessels were used as the recipient vessels.
  Interventions: Procedure: Recipient vessel selected for microanastomosis

INTERVENTIONS:
Procedure: Recipient vessel selected for microanastomosis — Free tissue flaps harvesting and microanastomosis were performed by the same surgeon and in a similar way in both group. Postoperative course, and complications were recorded and analyzed.

SUMMARY:
The goal of this clinical trial is to compare the postoperative outcomes based on superficial temporal versus cervical recipient vessels for midface and scalp advanced oncologic defects using free tissue flap for reconstruction.

The main question it aims to answer is:

• Which recipient vessel is most suitable for performing microanastomosis using free flaps for advanced midface and scalp oncologic defect.

Participants will be undergo resection of advanced malignant tumors of the midface and scalp with subsequent oncological reconstruction using free tissue flap.

Researchers will compare two groups where those in whom superficial temporal vessels will be used as the recipient vessels (group A) and those in whom cervical vessels will be used as the recipient vessels (group B) to see if there is a recipient vessel who is most suitable for performing microanastomosis using free flaps for advanced midface and scalp oncologic defect.

DETAILED DESCRIPTION:
Advanced oncologic defects of the midface and scalp are a significant challenge to the reconstructive head neck surgeon, who must consider the need for midfacial projection, rehabilitation, and function restoration. Free flaps reconstruction in the midface and scalp region are the gold standard for advanced cases. There is no consensus in the literature on which recipient vessel is most suitable for performing microanastomosis using free flaps for advanced midface and scalp oncologic defect. The aim of this clinical trial is prospectively compare the results of microvascular flap reconstruction of midface and scalp advanced oncologic defects using superficial temporal versus cervical as recipient vessels. This is a parallel trial with permuted block randomization of patients who will be undergone a midface and scalp oncologic reconstruction with free tissue flap. Two groups will be analyzed: those in whom superficial temporal vessels will be used as the recipient vessels (group A) and those in whom cervical vessels will be used as the recipient vessels (group B). Allocation ratio will de 1:1 participants. Patient gender and age, cause and localization of the defect, flap choice for reconstruction, recipient vessels, intraoperative outcome, postoperative course, and complications were recorded and analyzed. Considering that this is a disease with rare staging, the calculated sample size was 26, but it will be increased by 30% (total of 34 participants who will be selected) since the death rate of these patients ranges from 8-25% A Fisher's exact test will be used to compare outcomes between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to subtotal, total, or extensive radical oncologic maxillectomy, or advanced scalp oncologic defect
* Complete medical records for at least 30 days after the intervention
* Patients eligible for microanastomosis in both cervical and superficial temporal recipient vessels

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Serious diseases (sepsis, renal and hepatic failure, severe cardiovascular diseases, chronic obstructive pulmonary disease);
* Patients with HIV (human immunodeficiency virus) with or without AIDS (acquired immunodeficiency syndrome);
* Patients with synchronous malignant neoplasms of the upper airway-digestive tract;
* Patients who died within a period of less than 30 days or who were lost to follow-up for the same period

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
To compare the overall flap survival rate after the microanastomosis | Participants were assessed twice a day for the first 10 days after the intervention and then weekly for 4 weeks.
  Adequate perfusion of the free tissue flap was assessed using Doppler flowmetry, flap bleeding time after puncture, color, texture and turgor. Both venous and arterial thrombosis were evaluated by these methods in order to detect whether there was any evidence of low or absence of vascular perfusion of the flap.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno A Sousa, MD, Principal Investigator — Brazilian National Cancer Institute
Locations (1):
- Brazilian National Cancer Institute, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Awwad L, Obed D, Vogt PM, Kaltenborn A, Koenneker S. Superficial Temporal Recipient Vessels for Craniofacial Microvascular Free-Flaps. J Craniofac Surg. 2022 Sep 1;33(6):e652-e657. doi: 10.1097/SCS.0000000000008768. Epub 2022 Jul 22. PMID 35864586
- [Result] Mata Ribeiro L, Tsao CK, Hung YL, Chu CH, Lin LC, Lin MH, Peng C, Cheong DC, Hung SY, Liao CT. Venous Size Discrepancy Is a Critical Factor When Using Superficial Temporal Vessels as Recipient Vessels for Free Flaps. J Reconstr Microsurg. 2022 Oct;38(8):654-663. doi: 10.1055/s-0042-1743165. Epub 2022 Feb 25. PMID 35213928
- [Result] Sudirman SR, Shih HS, Chen JC, Feng KM, Jeng SF. Superficial temporal vessels, both anterograde and retrograde limbs, are viable recipient vessels for recurrent head and neck reconstruction in patients with frozen neck. Head Neck. 2019 Oct;41(10):3618-3623. doi: 10.1002/hed.25886. Epub 2019 Jul 26. PMID 31347733
- [Result] Mattine S, Payne KFB. The evolving role of the superficial temporal vessels as anastomotic recipients in challenging microvascular reconstruction of the upper two-thirds of the face. J Plast Reconstr Aesthet Surg. 2022 Sep;75(9):3330-3339. doi: 10.1016/j.bjps.2022.04.089. Epub 2022 May 2. PMID 35710778